CLINICAL TRIAL: NCT00276497
Title: Role of Pioglitazone in Preventing Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.V. Hospital for Diabetes (Other)
Collaborators: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDPP2
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Diabetes
Keywords: Impaired glucose tolerance; Intervention; Prevention
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pioglitazone

SUMMARY:
A three year prospective, double blinded, placebo controlled, randomized clinical trial in impaired glucose tolerance (IGT) subjects to study the effect of pioglitazone in preventing the conversion to Diabetes.

DETAILED DESCRIPTION:
A randomized controlled study was designed to find out whether pioglitazone will prevent the conversion to diabetes in subjects who are non obese and with impaired glucose tolerance.

It is a double blind prospective study for 3 years. The study was started in October 2003 and randomization was completed in May 2005. A total of 6643 subjects were screened and 406 were randomized either to pioglitazone or placebo(investigator blinded-groups assigned A and B). At randomisation subjects were given standard advice on diet,exercise and benefits of life style modifications.

Subjects both male and female, aged between 35 and 55 years, with no known history of diabetes, willing and available for a 3 year study alone were screened. Pregnant women, subjects with major illness such as cancer, hepatic or cardiac diseases and on transferable jobs were excluded from the study. The initial dose of tablet was 15mg o.d. which was titrated after a month to 30 mg o.d. in subjects who did not show any adverse events.

The subjects will be undergoing annual reviews with a repeat OGTT, for 3 years. An interim review at every six months is also being done. Proforma containing details of anthropometry, occupation, physical activity, dietary habits, details of medications, regularity of treatment will be done at each interview.

The main expected outcomes of the study will be a reduction in conversion of IGT to diabetes and benefits of the drug on anthropometric variables and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age 35 - 55 years
* No known history of diabetes
* Willing and available for a 3 years study

Exclusion Criteria:

* Pregnant women
* Subjects with major illness such as cancer, hepatic or cardiac diseases
* Transferable jobs

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2003-10; Study Completion 2008-05

PRIMARY OUTCOMES:
Reduction in conversion of IGT to diabetes

SECONDARY OUTCOMES:
benefits of the drug on anthropometric variables and biochemical parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ambady Ramachandran, MD,PhD,DSc, Principal Investigator — India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes hospitals, 28, Marshall's Road, Egmore, Chennai-600 008. India

REFERENCES:
- [Result] Ramachandran A, Snehalatha C, Mary S, Selvam S, Kumar CK, Seeli AC, Shetty AS. Pioglitazone does not enhance the effectiveness of lifestyle modification in preventing conversion of impaired glucose tolerance to diabetes in Asian Indians: results of the Indian Diabetes Prevention Programme-2 (IDPP-2). Diabetologia. 2009 Jun;52(6):1019-26. doi: 10.1007/s00125-009-1315-x. Epub 2009 Mar 10. PMID 19277602
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751